CLINICAL TRIAL: NCT01083277
Title: Variable Ventilation During Acute Respiratory Failure
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Boston Medical Center (Other)
Collaborators: Wallace H. Coulter Foundation (Other)
Responsible Party: Principal Investigator, Allan J. Walkey, BMC Attending Physician, Boston Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Device Feasibility
Other Study IDs: H-27864
Record Dates: First submitted 2009-09-18; First posted 2010-03-09 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Acute Respiratory Failure
Keywords: oxygenation; ventilation; tidal volume; patterns of breathing; variable ventilation; mechanical ventilation
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- variable ventilation (Experimental): A novel means of conducting mechanical ventilation that involves an approximately 40% variation in tidal volume around a set mean tidal volume
  Interventions: Device: variable ventilation
- conventional ventilation (Other): This is the control arm of the study, in which tidal volume will be set as the patient's baseline tidal volume prior to study entry and will not vary.
  Interventions: Other: Conventional ventilation

INTERVENTIONS:
Device: variable ventilation — In variable ventilation, the tidal volume on the Puritan-Bennett 840 ventilator will be randomly varied by 40% on a breath-by-breath basis around a pre-set mean, using the variable ventilation software developed by Dr. Bela Suki and Dr. Arnab Majumdar. In conventional ventilation, the tidal volume on the Puritan-Bennett 840 ventilator will be set to equal the mean tidal volume used in variable ventilation and does not vary.
  Arms: variable ventilation
Other: Conventional ventilation — tidal volume will be set as the patient's baseline tidal volume prior to study entry and will not vary.
  Arms: conventional ventilation

SUMMARY:
Acute respiratory failure requiring support with mechanical ventilation occurs with an incidence of 77-100 per 100,000 person-years and accounts for half of all patients admitted to the intensive care unit. Major causes of acute respiratory failure include pneumonia, asthma, emphysema, and acute lung injury. These causes of acute respiratory failure may result in partial lung collapse (atelectasis), and airway narrowing (bronchoconstriction)that result in decreased oxygen levels requiring support with the ventilator. The prolonged inactivity in the supine position associated with mechanical ventilation can further result in atelectasis requiring increased oxygen supplementation through the ventilator.

The current standard of care in acute respiratory failure is a strategy of mechanical ventilation using a single lung volume delivered repeatedly. However, the current standard mechanical ventilation strategy is not consistent with the variability in respiration of healthy humans and has been shown to contribute to increased lung injury in some studies. The mortality associated with acute respiratory failure is high, 30-40%. Thus, improvements in mechanical ventilation strategies that improve oxygen levels and potentially decrease further lung injury delivered by the ventilator are warranted.

Recent studies by BU Professor Bela Suki and others in humans and animals with acute lung injury, bronchoconstriction, and atelectasis have shown that varying the lung volumes delivered by a ventilator significantly decreases biomarkers of lung injury, improves lung mechanics, and increases oxygenation when compared to identical mean volumes of conventional, monotonous low lung volume ventilation.

Therefore, we propose a first-in-human, Phase I study to evaluate the safety of this novel mode of ventilation, Variable Ventilation, during acute respiratory failure

ELIGIBILITY:
Inclusion criteria

1. Age > or equal to 18
2. Requires mechanical ventilation using a volume-controlled mode.
3. Admitted to Boston Medical Center Surgical, Medical, or Coronary Intensive Care Unit
4. Evidence of impaired oxygenation on mechanical ventilator defined by PaO2/FiO2 ratio less than 350 (corresponding to an A-a gradient of approximately 100) or SatO2/FiO2 ratio less than 358 (requiring O2 saturation less than or equal to 97%).
5. Meets "Clinical Stability Criteria" (on maximum of one vasopressor medication) for at least one hour prior to start of study protocol:

5a. Hemodynamically stable: mean arterial pressure greater than 60 mmHg, heart rate greater than 50 and less than 130 bpm 5b. Respiratory system stable: Respiratory rate less than 35 bpm, O2 saturation greater than 88%, peak pressure on ventilator less than 40 cm H20, FiO2 not greater than 0.80, PEEP level not greater than 12.5 cm H2O, requires suctioning less than once hourly.

5c. Acid-base stability: pH greater than 7.2 and less than 7.55 5d. Neurologic system stable: No agitation as defined by a Riker SAS Score between 2 (very sedated) and 4 (calm and cooperative) 6. Assent of primary ICU care team

Exclusion Criteria

1. Do not resuscitate order
2. Increased intracranial pressure
3. Pregnancy (urine pregnancy test for all women of child-bearing age)
4. Planned transport out of ICU during planned study protocol
5. Coagulopathy (INR > 2.0 or PTT > 50)
6. Severe thrombocytopenia (platelets < 20,000)
7. Patients receiving medications meant to increase oxygenation such as inhaled nitric oxide, inhaled prostacyclin, intravenous prostacyclin, and intravenous treprostinil
8. Any patient receiving a medication that is not consistent with FDA-approved labeling
9. A change in the Riker SAS during the study protocol that results in a Riker SAS score of 1: "Unarousable" (minimal or no response to noxious stimuli, does not communicate or follow commands) or 5: "Agitation" (anxious or physically agitated, calms to verbal instructions) for a duration of greater than 15 minutes
10. A Riker SAS of 6: "Very agitated" (requiring restraint and frequent verbal reminding of limits, biting ETT) or higher will result in immediate study discontinuation for the individual participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2012-09; Primary Completion 2016-07 (Actual); Study Completion 2016-12-23 (Actual)

PRIMARY OUTCOMES:
The occurrence of adverse events in the use of variable ventilation versus conventional ventilation, including the loss of any of the following (1) hemodynamic stability, (2) respiratory stability,(3) acid-base stability, and (4) neurological stability. | Up to 24 hours after the end of the study period

SECONDARY OUTCOMES:
Oxygenation | 3 hours
  PaO2

OTHER OUTCOMES:
Biomarkers of lung injury | 3 hours
  IL6, IL8, IL1Ra, SP-D, sTNFaR I and II
Lung mechanics | 3 hours
  quasi static lung compliance, mean airway pressure, peak airway pressure, plateau pressure.
Sedatives | 3 hours
  need for increased sedative
PaCO2 | 3 hours

CONTACTS AND LOCATIONS:
Overall Officials: George T O'Connor, MD, Principal Investigator — Boston University
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No